CLINICAL TRIAL: NCT03484273
Title: Body Compression in Postural Tachycardia Syndrome (POTS): Effects on Orthostatic Tolerance
Brief Title: Hemodynamic Effects of Compression in POTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Satish Raj, Professor; Medical Director, Calgary Autonomic Investigation & Management Clinic, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REB17-2393
Record Dates: First submitted 2018-03-19; First posted 2018-03-30 (Actual); Results first posted 2021-05-12 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Postural Tachycardia Syndrome
Keywords: Tilt Table; Compression; Dysautonomia; POTS
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Autonomic Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: There will be 4 compression conditions based on strap configuration of the Lifewrap garment: full abdominal and lower extremity compression, abdominal only compression, lower extremity only compression and no compression. The order of these interventions will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Full Compression (Experimental): The LifeWrap compression garment will be fully secured with all straps.
  Interventions: Device: LifeWrap Compression Garment
- Abdominal and Pelvic Compression (Experimental): The Lifewrap compression garment abdominal, pelvic and upper thigh straps only will be secured.
  Interventions: Device: LifeWrap Compression Garment
- Lower Limb Compression (Experimental): The Lifewrap compression garment calf and ankle straps only will be secured.
  Interventions: Device: LifeWrap Compression Garment
- No Compression (No Intervention): None of the LifeWrap compression garment straps will be secured.

INTERVENTIONS:
Device: LifeWrap Compression Garment — Non-Pneumatic Anti-Shock (NASG) compression garment comprised of neoprene with velcro closures.
  Arms: Abdominal and Pelvic Compression; Full Compression; Lower Limb Compression

SUMMARY:
When an individual with Postural Tachycardia Syndrome (POTS) stands up, their heart rate increases significantly (>30BPM) and they may experience symptoms such as lightheadedness, dizziness, shortness of breath, nausea and mental confusion.

One commonly prescribed treatment for POTS is compression garments. Compression garments squeeze veins to help return blood back to the heart, which may decrease heart rate and symptoms on standing. However, there is little research about the effectiveness of compression in adults with POTS.

In this study, the investigators will use the Lifewrap garment, which compresses the abdomen, pelvis and lower extremities, to evaluate the effectiveness of compression in POTS. The investigators will use a head up tilt (HUT) which will simulate standing. The study participant will participate in 4x 10 minute HUTs wearing 4 different compression configurations:

1. full abdomen and lower extremity compression
2. abdominal only compression
3. leg only compression
4. No compression

The investigators hypothesize that with full compression, the participant's heart rate increase from lying down to upright will be lower than when they are not wearing any compression. The investigators will also ask the participant about their symptoms when they are upright.

The results of this study could demonstrate the potential benefits of compression and what configuration is most effective. These findings could rapidly translate to the clinical setting, providing improved care.

DETAILED DESCRIPTION:
Postural Tachycardia Syndrome (POTS) is a chronic form of orthostatic intolerance marked by a significant and sustained increase in heart rate (HR) upon positional change from supine to standing (>30 beats/min [bpm]) in the absence of orthostatic hypotension (<20/10 mmHg decrease). Symptoms must be present for >6 months and other causes of orthostatic tachycardia must be ruled out. Individuals with POTS report orthostatic symptoms including palpitations, lightheadedness, and mental clouding, which improve on recumbence. The vast majority of individuals diagnosed with POTS are women age 13-50 years.

Upon standing, approximately 500 mL of blood immediately redistributes from the thorax down to the abdomen, buttocks and legs. This leads to sympathetic activation as the baroreceptors sense less pressure. In a healthy individual, HR initially increases 10-20 bpm, and the systolic blood pressure (BP) decreases by approximately 5 mmHg. However, in an individual with POTS, this compensatory mechanism is impaired and HR will increase by >30 bpm and remain at this elevated rate for the duration of standing. In some individuals with POTS, upon standing cerebral blood flow velocity decreases. In other individuals, oscillation of cerebral blood flow due to failure of cerebral autoregulatory mechanisms is observed.

Current treatment of POTS involves pharmacological and non-pharmacological intervention including salt and fluid loading, exercise, and physical countermanuevers. There are no approved medications for use in POTS and all use is off label. Compression garments are also often prescribed. Abdominal/lower extremity compression garments provide pressure to the blood vessels in the legs, thighs and abdomen which can minimize blood pooling and lead to improved blood return to the heart. One such garment is the Lifewrap Non-pneumatic AntiShock garment (NASG), indicated in post-partum hypovolemia.

A pediatric study (n=20) found that orthostatic tachycardia and symptoms were decreased during head up tilt (HUT), with the use of a different NASG compression garment vs. no compression. However, there is no data to validate the efficacy of compression in adults POTS, and also no data to determine which type of compression is most beneficial (e.g. lower leg only, abdomen only, combination).

The investigators hypothesize that the use of the Lifewrap NASG compression garment in a fully applied configuration will decrease orthostatic tachycardia and orthostatic symptoms during a 10 minute HUT vs. no compression garment. The investigators will complete a 4-way randomized crossover study of HUTs with compression applied by the LifeWrap NSAG in at attempt to demonstrate decreased orthostatic tachycardia and increased orthostatic tolerance in individuals with POTS. If successful, this study could provide needed evidence that compression in POTS is a successful non-pharmacological treatment modality, and as well, what type of compression is the most beneficial to patients with this syndrome. These findings could rapidly translate to the clinical setting and improve patient care.

The study participant will complete 4x 10min HUTs during a single study day. There will be 4 compression conditions based on strap configuration of the Lifewrap garment: (1) full abdominal and lower extremity compression, (2) abdominal only compression, (3) lower extremity only compression and (4) no compression. A pressure sensor will used to measure the magnitude of compression pressure applied. The study will be conducted on a tilt table in a human physiology research and procedure room. Each intervention phase in the protocol will involve a supine baseline assessment period of 10 minutes followed by a 10 min HUT (80 degrees). There will be a 20 min recovery periods between each HUT. The study will take approximately 4 hours.

The study participant will be instrumented in a fasting state and on an empty bladder. The investigators will apply skin electrodes to continuously monitor heart rate and record an ECG. BP will be monitored continuously using a finger volume clamp method (Nexfin, Edwards Lifesciences) and calibrated with intermittent brachial cuff measurements (Vital-Guard 450C Patient Care Monitor, IVY Medical). From the continuous BP waveform, the investigators can obtain an estimate of stroke volume, cardiac output, and systemic vascular resistance (Modelflow). Middle cerebral blood flow velocity will be assessed using transcranial doppler.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of Postural Tachycardia Syndrome (POTS)
* Age 18-60 years (we are an adult group and we do not see pediatric patients clinically and do not have appropriate pediatric expertise)
* Male and Female
* Able and willing to provide informed consent
* Ability to travel to Libin Cardiovascular Institute of Alberta Autonomic Testing Lab at the University of Calgary, Calgary, AB.

Exclusion Criteria:

* Overt cause for postural tachycardia, i.e., acute dehydration
* Participants with somatization or severe anxiety symptoms will be excluded (as they may not tolerated study procedures)
* Pregnant women
* Inability to tolerate compression garment for the duration of the study
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD, MSCI, Principal Investigator — University of Calgary
Locations (1):
- Unversity of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bourne KM, Sheldon RS, Hall J, Lloyd M, Kogut K, Sheikh N, Jorge J, Ng J, Exner DV, Tyberg JV, Raj SR. Compression Garment Reduces Orthostatic Tachycardia and Symptoms in Patients With Postural Orthostatic Tachycardia Syndrome. J Am Coll Cardiol. 2021 Jan 26;77(3):285-296. doi: 10.1016/j.jacc.2020.11.040. PMID 33478652

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomized cross-over trial. Participants were assigned to receive the 4 compressions interventions in a randomized order. There were a total of 24 potential sequence orders of the compression interventions.
Groups:
- 4 Compression Interventions in Randomized Order: Participants completed all 4 compression garment interventions in a random order. There were a total of 24 possible intervention orders. The 4 compression interventions were: Full Compression, Abdominal and Pelvic Compression, Lower Limb Compression and No Compression.
Period: Overall Study
Arm/Group | 4 Compression Interventions in Randomized Order
Started | 32 (This was a crossover trial. A total of 32 participants were enrolled in this study.)
Completed | 30 (This was a crossover trial. A total of 30 participants completed all 4 arms.)
Not Completed | 2
Not completed — Equipment Malfunction | 1
Not completed — Data excluded from analysis | 1

BASELINE CHARACTERISTICS:
Arm/Group | Full Compression
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 30
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24 (6)

OUTCOME MEASURES:

1. Primary Outcome: Orthostatic Heart Rate (HR) Change
Description: The primary outcome measure will be the magnitude of HR change from supine to HUT (max HR between 5-10 min of HUT) for each study arm.
Time Frame: Maximum HR between 5-10min HUT MINUS the baseline (pre-tilt) HR
Population: This was a crossover trial. A total of 30 participants were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Full Compression | Abdominal and Pelvic Compression | Lower Limb Compression | No Compression
Number analyzed (Participants) | 30 | 30 | 30 | 30
beats per minute | 23 (11) | 28 (11) | 34 (14) | 39 (18)
Statistical Analysis 1: Comparison: Full Compression vs Abdominal and Pelvic Compression vs Lower Limb Compression vs No Compression; Repeated Measured ANOVA was used to compare the 4 compression garment configurations; Test type: Superiority; p < 0.001, ANOVA; Repeated Measures ANOVA

2. Secondary Outcome: Maximum Upright Heart Rate
Description: The maximum heart rate during minutes 5-10 of each HUT. The maximum heart rate during each of the study arms will be compared.
Time Frame: During minutes 5-10 of the HUT
Population: This was a crossover trial. A total of 30 participants were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Full Compression | Abdominal and Pelvic Compression | Lower Limb Compression | No Compression
Number analyzed (Participants) | 30 | 30 | 30 | 30
beats per minute (bpm) | 92 (14) | 97 (15) | 103 (16) | 109 (19)
Statistical Analysis 1: Comparison: Full Compression vs Abdominal and Pelvic Compression vs Lower Limb Compression vs No Compression; Test type: Superiority; p < 0.001, Repeated Measures ANOVA

3. Secondary Outcome: Differences in Vanderbilt Orthostatic Symptom Score (VOSS) Symptom Rating
Description: Subjective symptom scoring as reported by participant during each study arm. The VOSS evaluates 9 symptoms on a 0 to 10 scale with 0 being no symptom to 10 being worst ever symptom. The total score ranges from 0-90, with a higher score being more severe symptoms.
  The 9 symptoms are mental clouding, blurred vision, shortness of breath, rapid heartbeat, tremulousness, chest discomfort, headache, lightheadedness, and nausea. The participant's VOSS score will be compared across the 4 arms of this study.
  The VOSS score has been previously used in multiple publications
Time Frame: After t=10 of the 10min HUT (or sooner if HUT has to be terminated early due to symptoms)
Population: This was a crossover trial. A total of 30 participants were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Compression | Abdominal and Pelvic Compression | Lower Limb Compression | No Compression
Number analyzed (Participants) | 30 | 30 | 30 | 30
units on a scale | 12 (10) | 15 (12) | 22 (17) | 26 (17)
Statistical Analysis 1: Comparison: Full Compression vs Abdominal and Pelvic Compression vs Lower Limb Compression vs No Compression; Test type: Superiority; p < 0.001, Repeated Measures ANOVA

4. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Change in continuous systolic blood pressure between supine and HUT during each study arm.
Time Frame: During the baseline before the HUT and the SBP correlating with the maximum HR during 5-10 min HUT, recorded at 1 min intervals.
Population: This was a crossover trial. A total of 29 participants were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Full Compression | Abdominal and Pelvic Compression | Lower Limb Compression | No Compression
Number analyzed (Participants) | 29 | 29 | 29 | 29
mmHg | -5 (7) | -7 (8) | -10 (10) | -10 (10)
Statistical Analysis 1: Comparison: Full Compression vs Abdominal and Pelvic Compression vs Lower Limb Compression vs No Compression; Test type: Superiority; p = 0.01, Repeated Measures ANOVA

5. Secondary Outcome: Changes in Stroke Volume
Description: Change in Stroke Volume from supine to HUT in each of the study arms.
Time Frame: During the baseline before the HUT and the SV correlating with the maximum HR during 5-10 min HUT, recorded at 1 min intervals.
Population: This was a crossover trial. A total of 29 participants were analyzed.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Full Compression | Abdominal and Pelvic Compression | Lower Limb Compression | No Compression
Number analyzed (Participants) | 29 | 29 | 29 | 29
mL | -22 (12) | -22 (12) | -33 (14) | -34 (11)
Statistical Analysis 1: Comparison: Full Compression vs Abdominal and Pelvic Compression vs Lower Limb Compression vs No Compression; Test type: Superiority; p < 0.001, Repeated Measures ANOVA

6. Secondary Outcome: Change in Cardiac Output (CO)
Description: Change in Cardiac Output from supine to HUT in each of the study arms.
Time Frame: During the baseline before the HUT and the CO correlating with the maximum HR during 5-10 min HUT, recorded at 1 min intervals.
Population: This was a crossover trial. A total of 29 participants were analyzed.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Full Compression | Abdominal and Pelvic Compression | Lower Limb Compression | No Compression
Number analyzed (Participants) | 29 | 29 | 29 | 29
L/min | 0.1 (0.7) | 0.3 (0.7) | -0.2 (1) | -0.2 (0.8)
Statistical Analysis 1: Comparison: Full Compression vs Abdominal and Pelvic Compression vs Lower Limb Compression vs No Compression; Test type: Superiority; p = 0.001, Repeated Measures ANOVA

7. Secondary Outcome: Change in Systemic Vascular Resistance (SVR)
Description: Change in Systemic Vascular Resistance from supine to HUT in each of the study arms.
Time Frame: During the baseline before the HUT and the SVRcorrelating with the maximum HR during 5-10 min HUT, recorded at 1min intervals.
Population: This was a crossover trial. A total of 29 participants were analyzed.
Measure: Mean (Standard Deviation); unit: dyne*s/cm^5
Arm/Group | Full Compression | Abdominal and Pelvic Compression | Lower Limb Compression | No Compression
Number analyzed (Participants) | 29 | 29 | 29 | 29
dyne*s/cm^5 | -31 (132) | -63 (152) | -22 (157) | 4.7 (145)
Statistical Analysis 1: Comparison: Full Compression vs Abdominal and Pelvic Compression vs Lower Limb Compression vs No Compression; Test type: Superiority; p = 0.04, Repeated Measures ANOVA

8. Secondary Outcome: Change in Cerebral Blood Flow Velocity (CBFV)
Description: Change in cerebral blood flow from supine to HUT in each of the study arms.
Time Frame: During the baseline before the HUT and the CBFV correlating with the maximum HR during 5-10 min HUT, recorded at 1 min intervals.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: This was a half day study and there was no ongoing follow up.
Arm/Group | Full Compression | Abdominal and Pelvic Compression | Lower Limb Compression | No Compression
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32

LIMITATIONS AND CAVEATS:
This was a proof of principle study. The garment used is not one that a typical patient would use in their day to day lives. The use of "real-world" garments requires further testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT03484273/Prot_SAP_000.pdf